CLINICAL TRIAL: NCT01034709
Title: Clinical Evaluation of the Artus® CMV RG PCR Test
Brief Title: Evaluation of the Artus® CMV PCR Test
Acronym: CMV
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: C09-CMV-001
Record Dates: First submitted 2009-12-15; First posted 2009-12-17 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Cytomegalovirus Infections
Keywords: Cytomegalovirus; CMV
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extracted DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Symptomatic: Subjects with a confirmed CMV viremia by the site's CMV-LDT as well as CMV symptoms
- Asymptomatic: Subjects who must have been serologically positive for CMV IgG prior to transplantation and do not have any CMV symptoms

SUMMARY:
Subjects with symptomatic CMV infection, who are enrolled in this clinical study, will be monitored during antiviral therapy.

DETAILED DESCRIPTION:
The human Cytomegalovirus (CMV) is found in blood, tissues and nearly all secretory fluids of infected persons. Transmission can be oral, sexual, via blood transfusion, organ transplantation, intrauterine, or perinatal. Infection with CMV preadolescence frequently leads to an asymptomatic infection followed by a lifelong persistence of the virus in the body. Infection post adolescence typically leads to symptoms that resemble those of mononucleosis (e.g., fever, fatigue, hepatitis, etc.) In contrast, CMV infections in immune compromised patients can be life threatening. A major cause of virus-associated morbidity and mortality in solid organ transplantation patients is illness caused by CMV (i.e., CMV syndrome or CMV disease).

The risk of progressing to CMV disease post-transplant is strongly correlated with the serological status of the donor (D) and recipient (R); the highest risk group is R-/D+. Patients at risk for CMV disease can be managed either preemptively (i.e., patients are only treated with antiviral agents after evidence of CMV infection arises), or prophylactically (i.e., all patients are treated with antiviral agents regardless of CMV infection status). Monitoring of the CMV viral load of transplant patients during antiviral therapy provides an effective aid in the management of patients with CMV disease. The artus® CMV RG PCR test is a nucleic acid amplification-based assay for the quantitation of CMV DNA using PCR in the Rotor-Gene™ 6000 Instrument (also known as Rotor-Gene Q) with software version 2.0.2.3 or higher. In the present study the artus CMV RG PCR test result will be evaluated for its ability to safely and effectively monitor transplant patients during antiviral therapy and will be compared to the COBAS® AmpliPrep/COBAS® TaqMan® CMV Test

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have had a kidney transplant.
2. Subjects that present at a hospital, clinic or physicians office for post-transplantation care.
3. Subjects must be 18 years of age or older.
4. Subjects providing informed consent.
5. Subjects must have a CMV infection as demonstrated by a positive result by the site's CMV-PCR-Laboratory Developed Test (CMV-PCR-LDT)
6. Subjects must be candidates for, and will be treated with ganciclovir and/or valganciclovir antiviral therapy.

Exclusion Criteria:

1. Subjects wherein the HIV status is positive.
2. Specimens with less than 1.0 ml EDTA plasma for artus testing.
3. Subjects from whom samples were collected, handled and/or stored inappropriately and/or determined to be unsatisfactory for processing/testing with the artus CMV RG PCR test (for which an explanation is provided in the case of subject exclusion).

   EDTA plasma specimens that have been stored inappropriately which include the following storage conditions: whole blood that has been frozen; whole blood processed for plasma more than 24 hours after collection; plasma stored at room temperature for more than 24 hours or 4C for more than 5 days at -20C for more than 6 months; frozen plasma with more than two freeze thaw cycles;

   Extracted nucleic acid that has been stored inappropriately which include the following storage conditions: extracted DNA stored for more than 5 days at -20C, or longer than six months at -20C; frozen nucleic acid with more than two freeze/thaw cycles.
4. Specimens that have been stored inappropriately for testing with that test used by the site to demonstrate a CMV infection. (A site specific memo will be provided to QIAGEN on appropriate specimen storage conditions.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes subjects that have received a kidney transplant, and that are hospitalized or that present to a hospital, clinic or physicians office for post-transplantation care and will be treated with ganciclovir and/or valganciclovir for symptomatic CMV infection.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2009-12; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California - Los Angeles, Los Angeles, California
  - University of Miami, Miami, Florida
  - LifeLink Health Care Institute, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana

REFERENCES:
- [Background] Patel R, Paya CV. Infections in solid-organ transplant recipients. Clin Microbiol Rev. 1997 Jan;10(1):86-124. doi: 10.1128/CMR.10.1.86. PMID 8993860
- [Background] Humar A, Michaels M; AST ID Working Group on Infectious Disease Monitoring. American Society of Transplantation recommendations for screening, monitoring and reporting of infectious complications in immunosuppression trials in recipients of organ transplantation. Am J Transplant. 2006 Feb;6(2):262-74. doi: 10.1111/j.1600-6143.2005.01207.x. PMID 16426310
- [Background] Greanya ED, Partovi N, Yoshida EM, Shapiro RJ, Levy RD, Sherlock CH, Stephens GM. The role of the cytomegalovirus antigenemia assay in the detection and prevention of cytomegalovirus syndrome and disease in solid organ transplant recipients: A review of the British Columbia experience. Can J Infect Dis Med Microbiol. 2005 Nov;16(6):335-41. doi: 10.1155/2005/679386. PMID 18159516
- [Background] Kanj SS, Sharara AI, Clavien PA, Hamilton JD. Cytomegalovirus infection following liver transplantation: review of the literature. Clin Infect Dis. 1996 Mar;22(3):537-49. doi: 10.1093/clinids/22.3.537. PMID 8852975
- [Background] Paya C, Humar A, Dominguez E, Washburn K, Blumberg E, Alexander B, Freeman R, Heaton N, Pescovitz MD; Valganciclovir Solid Organ Transplant Study Group. Efficacy and safety of valganciclovir vs. oral ganciclovir for prevention of cytomegalovirus disease in solid organ transplant recipients. Am J Transplant. 2004 Apr;4(4):611-20. doi: 10.1111/j.1600-6143.2004.00382.x. PMID 15023154
- [Background] Sia IG, Wilson JA, Groettum CM, Espy MJ, Smith TF, Paya CV. Cytomegalovirus (CMV) DNA load predicts relapsing CMV infection after solid organ transplantation. J Infect Dis. 2000 Feb;181(2):717-20. doi: 10.1086/315242. PMID 10669361
- [Background] Singh N. Cytomegalovirus infection in solid organ transplant recipients: new challenges and their implications for preventive strategies. J Clin Virol. 2006 Apr;35(4):474-7. doi: 10.1016/j.jcv.2005.10.014. Epub 2006 Jan 6. PMID 16406798
- [Background] Hadaya K, Wunderli W, Deffernez C, Martin PY, Mentha G, Binet I, Perrin L, Kaiser L. Monitoring of cytomegalovirus infection in solid-organ transplant recipients by an ultrasensitive plasma PCR assay. J Clin Microbiol. 2003 Aug;41(8):3757-64. doi: 10.1128/JCM.41.8.3757-3764.2003. PMID 12904387
- [Background] Humar A, Gregson D, Caliendo AM, McGeer A, Malkan G, Krajden M, Corey P, Greig P, Walmsley S, Levy G, Mazzulli T. Clinical utility of quantitative cytomegalovirus viral load determination for predicting cytomegalovirus disease in liver transplant recipients. Transplantation. 1999 Nov 15;68(9):1305-11. doi: 10.1097/00007890-199911150-00015. PMID 10573068
- [Background] Humar A, Siegal D, Moussa G, Kumar D. A prospective assessment of valganciclovir for the treatment of cytomegalovirus infection and disease in transplant recipients. J Infect Dis. 2005 Oct 1;192(7):1154-7. doi: 10.1086/444398. Epub 2005 Aug 23. PMID 16136456
- [Background] Piiparinen H, Helantera I, Lappalainen M, Suni J, Koskinen P, Gronhagen-Riska C, Lautenschlager I. Quantitative PCR in the diagnosis of CMV infection and in the monitoring of viral load during the antiviral treatment in renal transplant patients. J Med Virol. 2005 Jul;76(3):367-72. doi: 10.1002/jmv.20367. PMID 15902704
- See also: Organ Procurement and Transplant Network — http://optn.transplant.hrsa.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Symptomatic: Subjects with a confirmed CMV viremia by the site's CMV-LDT
- Asymptomatic: Subjects who are serologically negative for CMV IgG prior to transplantation and do not have any CMV symptoms
Period: Overall Study
Arm/Group | Symptomatic | Asymptomatic
Started | 53 | 58
Completed | 44 | 42
Not Completed | 9 | 16
Not completed — Protocol Violation | 9 | 16

BASELINE CHARACTERISTICS:
Population: Age, gender, and race/ethnicity data was not collected for the Asymptomatic arm of this study.
Groups:
- Asymptomatic: Subjects who are serologically negative for CMV IgG
- Total: Total of all reporting groups
Arm/Group | Symptomatic | Asymptomatic | Total
Number analyzed (Participants) | 44 | 0 | 44
Age, Continuous [Mean (Full Range); unit: years] | 49 [22 to 72] |  | 49 [22 to 72]
Gender [Number; unit: participants]
  Female | 19 |  | 19
  Male | 25 |  | 25
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6 |  | 6
  Black or African American/ Not Hispanic or Latino | 14 |  | 14
  Black/Hispanic or Latino | 1 |  | 1
  White/Hispanic or Latino | 8 |  | 8
  White/Not Hispanic or Latino | 9 |  | 9
  Other | 1 |  | 1
  Native Hawaiian/Other Pacific Islander | 1 |  | 1
  Hispanic/Latino | 4 |  | 4
Region of Enrollment [Number; unit: participants]
  United States | 44 |  | 44

OUTCOME MEASURES:

1. Primary Outcome: a) CMV Viral Load
Description: The CMV viral load was measured by both the artus CMV RG PCR test and the COBAS® AmpliPrep/COBAS® TaqMan® CMV Test at the investigational sites and then the percent agreement between the two tests was determined.
Time Frame: 3 months
Measure: Number; unit: percentage of agreement
Arm/Group | Symptomatic | Asymptomatic
Number analyzed (Participants) | 44 | 42
percentage of agreement
  Not Detected | 100 | 97.6
  LOQ IU/ml | 86.36 | NA — No participants with detectable level in this group
  500 IU/ml | 95.45 | NA — No participants with detectable level in this group
  1000 IU/ml | 90.91 | NA — No participants with detectable level in this group

ADVERSE EVENTS:
Time Frame: At time of blood collection.
Arm/Group | Symptomatic | Asymptomatic
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/42
Other Adverse Events (participants affected / at risk) | 0/44 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No